CLINICAL TRIAL: NCT07183501
Title: Combined Hystroscopic and Laparoscopic Repair of CS Scar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Muhammad Rageh, Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Managment of CS scar disorder
Record Dates: First submitted 2025-09-05; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section Complications; Abnormal Uterine Bleeding
Keywords: Cesarean Section; niche; CSD
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with symptomatic uterine niche (Experimental)
  Interventions: Procedure: Combined hystroscopic and laparoscopic repair

INTERVENTIONS:
Procedure: Combined hystroscopic and laparoscopic repair — Hystroscopic isthmoplasty will be done first to ensure removal of chronically inflamed Unhealthy edges of niche, then laparoscopic exison of scar will be dine, followed by repair of the defect

SUMMARY:
Combined hystroscopic and laparoscopic repair of symptomatic uterine Niche as new technique to maximize resolution of symptoms after niche repair with concomitant increase in RMT

ELIGIBILITY:
Inclusion Criteria:

* symptomatic uterine Niche :postmenstrual spotting

Exclusion Criteria:

* contraindications for endoscopy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
change in Residual Myometrial Thickness | 3 months
  in mm

SECONDARY OUTCOMES:
Number of patients complete resolution of symptoms | 3 months
  dissappearance of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, women health hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided